CLINICAL TRIAL: NCT05112380
Title: Elaboration of an External Rotators Fatigue Test With an XCo
Brief Title: Fatigue Test With an XCo
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Physiotherapist, University of Liege
Other Study IDs: Fatigue XCo
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sedentary adults: * Do not practice overhead sport
  * No pain or history of shoulder pain
  Interventions: Other: Performing Xco endurance test
- Overhead athletes: * Practice an overhead sport at least five hours a week
  * No pain or history of shoulder pain
  Interventions: Other: Performing Xco endurance test

INTERVENTIONS:
Other: Performing Xco endurance test — The subjects will perform the test two times, with 7-10 days between the two sessions

SUMMARY:
The reliability of the Xco endurance test will be assessed in sedentary adults and in overhead athletes. The experimentation will be divided into two sessions. During the sessions, the impact of the test on rotators strength and throwing performance will be explored.

DETAILED DESCRIPTION:
At first, the reliability of the Xco endurance test will be assessed in sedentary adults. Then, the reliability of the test will be assessed in overhead athletes. The experimentation will include two sessions. During those sessions, the impact of fatigue (induced by the test) on rotator cuff muscles strength and on functional test performance (Single Arm Medicine Ball Throw) will be assessed. A time of 7 to 10 days will be provided between the two sessions.

To perform the XCo endurance test, the participant will be seated on a chair, arm at 90° of abduction (in frontal plane), elbow flexed at 90 degrees and positioned on a wooden support. From a 90 degrees of abduction and a neutral position of rotation, the participants will be asked to realise an external rotation movement of 90 degrees and then to go back to the starting position as many times as possible at a speed of 140 bpm. Mechanical stops (the wall and an adjustable height table) will be added to make sure that the participants respected the entire range of motion. After adjusting the position, it will be asked to the participants to perform 2 repetitions of 5 movements at 140 bpm (in eccentric and concentric) to get familiar to the rhythm. Thirty seconds of rest will be provided between the 2 repetitions to avoid the appearance of fatigue before the test.

Then, the participants will begin the test. The objective of the test will be to perform the movement as long as possible. The test will be stopped if the volunteers is not able to maintain the rhythm or to do the movement anymore. The Modified Borg Scale will be used to be sure that each subject was really exhausted when the test was stopped. For that purpose, each of them will have to quantify their level of exhaustion on the scale (maximum score = 10) every 30 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Practice of an overhead sport at least 5 hours a week (overhead athletes group)
* Not practice an overhead sport (sedentary adults)

Exclusion Criteria:

* History of shoulder pain
* Shoulder pain

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population will be divided into two groups : sedentary adults and overhead athletes
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Time to exhaustion | 10 days
Shoulder rotators strength | 10 minutes
Distance reached with Single Arm Medicine Ball Throw | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Camille Tooth, Principal Investigator — ULiège
Locations (1):
- Université de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tooth C, Forthomme B, Croisier JL, Gofflot A, Bornheim S, Schwartz C. The Modified-Athletic Shoulder Test: Reliability and validity of a new on-field assessment tool. Phys Ther Sport. 2022 Nov;58:8-15. doi: 10.1016/j.ptsp.2022.08.003. Epub 2022 Aug 30. PMID 36088802